CLINICAL TRIAL: NCT05575921
Title: Diagnostic of Sleep Obstructive Apnea Syndrome in Children by Home Sleep Studies
Brief Title: Diagnostic of Sleep Obstructive Apnea Syndrome in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr. Iulia IOAN, MD PhD Associate Professor, Central Hospital, Nancy, France
Other Study IDs: 2022PI145-309
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Apnea, Obstructive Sleep
Keywords: Sleep apnea; Child; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — Children underwent at-home polysomnography in routine clinical practice. The exam is interpreted in 2 ways by the physician with sleep stages (PSG) and without sleep stages (PG). The data are retrospectively collected from the patient's recording

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) in children is a significant public health problem whose clinical diagnosis is not specific. The recording of sleep and breathing (polysomnography, PSG) is the reference exam. PSG consists in installing on the child's body electrodes necessary to determine the sleep stages and sensors used to determine the presence of respiratory events during sleep. At-home PSG, compared to hospital PSG, improves sleep quality. PSG is yet an anxious exam due to the multitude of electrodes and sensors. Ventilatory polygraphy (PG) consists of installing only respiratory detectors.

The objective of this study is to demonstrate that at-home PG has the same diagnostic value as at-home PSG.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome (OSAS) in children causes chronic hematosis disorders and sleep disruption that negatively impacts growth, neurocognitive performance, and cardiovascular and metabolic functions. Its high frequency makes it a major public health problem. The clinical elements for the diagnosis are not specific and the recording of sleep and breathing (polysomnography, PSG) is the reference exam (HAS Recommendations, 2012). PSG consists in installing on a child's body electroencephalogram (EEG), electrooculogram (EOG), and electromyogram (EMG) electrodes, necessary to determine the sleep stages and sleep-wake periods, and also the sensors used to determine the presence of respiratory events during sleep such as a nasal cannula, thoracoabdominal belts, oximetry, and actimetry. At-home PSG, compared to hospital PSG, improves sleep quality and diagnostic conditions. But the PSG remains a rather anxious exam for the child due to the multitude of electrodes and sensors. Ventilatory polygraphy (PG) consists of installing only the respiratory detectors (nasal cannula, thoracoabdominal belts, oximetry, and actimetry), without the EEG, EOG, and EMG electrodes. Several studies in the literature have compared these 2 exams, PSG and PG, for diagnosing OSAS in children with varied and sometimes contradictory results.

The hypothesis of the study is that the obstructive apnea-hypopnea index (OAHI, the number of apneas, and obstructive hypopneas per hour) obtained by at-home PSG and the OAHI obtained by at-home PG are not different. For this, the sleep physician will analyze the sleep recording performed at home in routine clinical practice, in 2 ways: 1) by determining the sleep stages and computing OAHI per hour of sleep; 2) by removing EEG, EOG, and EMG signals and computing OAHI over the duration of the sleep estimated by the physician according to child's behavior during sleep (movements, artifacts) as in PG.

The main objective of this study is to demonstrate that at-home PG has the same diagnostic value as at-home PSG, i.e. OAHI obtained by at-home PG is similar to OAHI obtained by at-home PSG. The second objective is to determine the faisability in terms of the percentage of interpretable exams of at-home PSG.

ELIGIBILITY:
Inclusion Criteria:

* Data from at-home PSG retrospectively collected from the hospital recording of children who underwent an exam during the period October 2020 to March 2021

Exclusion Criteria:

-

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Data from at-home PSG retrospectively collected from the hospital recording of children who underwent an exam during the period October 2020 to March 2021
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
At-home PG has the same diagnostic value than at-home PSG | One night
  OAHI obtained by at-home PG is similar to OAHI obtained by at-home PSG

SECONDARY OUTCOMES:
At-home PSG faisability | 1 hour
  To determine the faisability in terms of the percentage of interpretable exam for at-home PSG

REFERENCES:
- [Result] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Result] Mitchell RB, Pereira KD, Friedman NR. Sleep-disordered breathing in children: survey of current practice. Laryngoscope. 2006 Jun;116(6):956-8. doi: 10.1097/01.MLG.0000216413.22408.FD. PMID 16735907
- [Result] Masoud AI, Patwari PP, Adavadkar PA, Arantes H, Park C, Carley DW. Validation of the MediByte Portable Monitor for the Diagnosis of Sleep Apnea in Pediatric Patients. J Clin Sleep Med. 2019 May 15;15(5):733-742. doi: 10.5664/jcsm.7764. PMID 31053204
- [Result] Lesser DJ, Haddad GG, Bush RA, Pian MS. The utility of a portable recording device for screening of obstructive sleep apnea in obese adolescents. J Clin Sleep Med. 2012 Jun 15;8(3):271-7. doi: 10.5664/jcsm.1912. PMID 22701384
- [Result] Massicotte C, Al-Saleh S, Witmans M, Narang I. The utility of a portable sleep monitor to diagnose sleep-disordered breathing in a pediatric population. Can Respir J. 2014 Jan-Feb;21(1):31-5. doi: 10.1155/2014/271061. Epub 2013 Sep 30. PMID 24083303